CLINICAL TRIAL: NCT06433115
Title: Effects of Lean Beef Consumption on Cardiometabolic Health and Gut Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jaapna Dhillon, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2097458; 2097458 (Other: University of Missouri)
Record Dates: First submitted 2024-04-29; First posted 2024-05-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Diet Intervention
MeSH Terms: interventions — Meat Substitutes

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lean (≥90%) Grass-Fed Beef (Experimental): The quantity of beef will be adjusted or normalized based on their individual energy requirements. The specified amount will be 4 oz. per day or 28 ounces per week for participants with an energy requirement of 2000 kcal. Participants will consume meals for six weeks.
  Interventions: Other: Lean (≥90%) Grass-Fed Beef
- Lean (≥90%) Grain-Fed Beef (Experimental): The quantity of beef will be adjusted or normalized based on their individual energy requirements. The specified amount will be 4 oz. per day or 28 ounces per week for participants with an energy requirement of 2000 kcal. Participants will consume meals for six weeks.
  Interventions: Other: Lean (≥90%) Grain-Fed Beef
- Plant-Based Meat (Active Comparator): Plant-based meat (beyond meat product) would be macronutrient matched to the same quantities of meat prescribed for a given energy level. Participants will consume meals for six weeks.
  Interventions: Other: Plant-Based Meat

INTERVENTIONS:
Other: Lean (≥90%) Grass-Fed Beef — The specified amount will be 4 oz. per day or 28 ounces per week for participants with an energy requirement of 2000 kcal.
  Arms: Lean (≥90%) Grass-Fed Beef
Other: Lean (≥90%) Grain-Fed Beef — The specified amount will be 4 oz. per day or 28 ounces per week for participants with an energy requirement of 2000 kcal.
  Arms: Lean (≥90%) Grain-Fed Beef
Other: Plant-Based Meat — Plant-based meat would be macronutrient matched to the same quantities of meat prescribed for a given energy level.
  Arms: Plant-Based Meat

SUMMARY:
This study is investigating the benefits of lean beef consumption on cardiometabolic health and gut microbiome.

DETAILED DESCRIPTION:
The study is a 6-wk randomized, controlled, and parallel arm clinical trial. Participants will be randomized to consume either lean grain-fed beef, lean grass-fed beef, or plant-based meat for 6 weeks. Outcomes assessed will include metabolic, inflammatory, and gut microbiome markers.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years of age
* BMI: 18-35 kg/m2
* Willingness to consume study foods.
* Willing to comply with study protocol.
* Consistent diet and activity patterns for 4 weeks
* Weight stable (≤5 kg change over the last 3 months)
* Non-smoker >1 year or more

Exclusion Criteria:

* Allergies to foods provided in the study
* Diabetes
* Gastrointestinal disease and/or bariatric surgery
* Uncontrolled hypertension and blood pressure ≥ 180/110
* Illicit drug use
* Recent consumption of antibiotics or probiotics
* Recent start of medications that affect metabolism or appetite.
* Recent blood donation
* Drug therapy for coronary artery disease, peripheral artery disease, congestive - heart failure, or dyslipidemia
* Pregnant or lactating individuals
* Taste or smell disorders
* High consumers of red meat or plant-based meat (≥ 4 times/week)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
LDL-C concentrations | Baseline, week 6
  Lipid profile
Interleukin-6 concentrations | Baseline, week 6
  Inflammatory marker
Gut microbial alpha-diversity | Baseline, week 6
  Assessed via16S rRNA sequencing

SECONDARY OUTCOMES:
HDL-C concentrations | Baseline, week 6
  Lipid profile
Total cholesterol concentrations | Baseline, week 6
  Lipid profile
Triglyceride concentrations | Baseline, week 6
  Lipid profile
Gut microbiome abundance | Baseline, week 6
  16S rRNA sequencing
LPS-binding protein concentration | Baseline, week 6
  Intestinal permeability marker
Glucose concentrations | Baseline, week 6
  Blood Glucose
Insulin concentrations | Baseline, week 6
  Insulin
Body mass | Baseline, week 3, and week 6
  Measured in kg
Fat mass | Baseline, week 3, and week 6
  Fat mass
Fat-free mass | Baseline, week 3, and week 6
  Fat-free mass
Waist circumference | Baseline, week 3, and week 6
  Waist circumference
Hip circumference | Baseline, week 3, and week 6
  Hip Circumference
Thigh circumference | Baseline, week 3, and week 6
  Thigh Circumference
24 hour appetite ratings | Baseline, week 6
  24-hour appetite ratings assessed on VAS
Physical activity scores | Baseline, week 6
  Activity assessment using Actigraphs
Total hours of sleep | Baseline, week 6
  Sleep diary
Palatability rating of foods | Baseline, week 3, week 6
  Hedonic general labelled magnitude scale (gLMS)
Acceptance rating of foods | Baseline, week 3, week 6
  9-point food action rating scale
Taste and flavor intensity ratings of foods | Baseline
  Sensory intensity scales
Gene expression levels | Baseline, week 6
  Transcriptomics analyses
Inflammatory marker concentrations | Baseline, week 6
  Inflammatory markers
Healthy eating index score | Baseline, week 6
  NCI diet history questionnaire

OTHER OUTCOMES:
Metabolite intensities | Baseline, week 6
  Untargeted and targeted metabolomics
Nutrient intakes | Baseline, week 3, week 6
  24 hours dietary recall

CONTACTS AND LOCATIONS:
Overall Officials: Jaapna Dhillon, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported here after deidentification (ie; text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be deposited in online repositories